CLINICAL TRIAL: NCT06570096
Title: Premixed Versus Sequential Injections of Lidocaine and Bupivacaine for Supraclavicular Brachial Plexus Block in Patients Undergoing Arteriovenous Fistula Creation: A Randomized Clinical Trial
Brief Title: Premixed vs Sequential Injections of Lidocaine and Bupivacaine for Supraclavicular Brachial Plexus Block in Patients Undergoing Arteriovenous Fistula Creation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR746/7/2024
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Premixed; Sequential; Lidocaine; Bupivacaine; Supraclavicular Brachial Plexus Block; Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential Injections group (Experimental): Patients will receive 10 ml of lidocaine 2% then 10 ml of bupivacaine 0.5% with a delay of 120s between injections.
  Interventions: Drug: Lidocaine 2% then bupivacaine 0.5%
- Premixed Injections group (Active Comparator): Patients will receive 20 ml of freshly prepared mixtures of 10 ml of lidocaine 2% and 10 ml of bupivacaine 0.5%
  Interventions: Drug: Lidocaine 2% and bupivacaine 0.5%

INTERVENTIONS:
Drug: Lidocaine 2% then bupivacaine 0.5% — Patients will receive 10 ml of lidocaine 2% then 10 ml of bupivacaine 0.5% with a delay of 120s between injections.
  Arms: Sequential Injections group
Drug: Lidocaine 2% and bupivacaine 0.5% — Patients will receive 20 ml of freshly prepared mixtures of 10 ml of lidocaine 2% and 10 ml of bupivacaine 0.5%.
  Arms: Premixed Injections group

SUMMARY:
This study aims to compare premixed and sequential injections of lidocaine and bupivacaine for supraclavicular brachial plexus block in patients undergoing arteriovenous fistula creation.

DETAILED DESCRIPTION:
Hemodialysis is the common treatment for end-stage renal disease (ESRD) condition which improves quality of life and survival rate for this group of patients. Arteriovenous fistula (AVF) creation is the vascular access technique that provides long-term vascular access for hemodialysis patients.

Ultrasound-guided supraclavicular brachial plexus block (SCBPB) is a widely accepted and effective technique for AVF creation procedures. It provides analgesia, sympathetic blockade, optimal surgical conditions, and adequate duration of postoperative block that prevents arterial spasm and graft thrombosis. It offers higher blood flow in the radial artery and arteriovenous fistula than is achieved with infiltration anesthesia.

Lipid-soluble local anesthetics (LA) such as ropivacaine and bupivacaine are generally more potent and have a significantly longer duration of action as well as a more prolonged onset of action compared to intermediate-potency drugs such as lignocaine, mepivacaine, and prilocaine. A combination of two LAs is often used in regional blocks to utilize the different clinical properties of the drugs to achieve a faster onset and longer block duration.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status III.
* Undergoing arteriovenous Fistula creation.

Exclusion Criteria:

* Allergy to local anesthetics.
* Body mass index (BMI) ≥ 35 kg/m2.
* Preoperative neurological deficit.
* Neuromuscular disorder.
* Psychiatric disorder.
* Coagulation disorder.
* Congestive heart failure.
* Pregnancy.
* Infection at the site of block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-24 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-03-16 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a complete four-nerve sensory block | With in 10 minutes intraoperatively
  Percentage of participants with a complete four-nerve sensory block at 10 minutes will be recorded.

SECONDARY OUTCOMES:
Time of onset of sensory block | Intraoperatively
  Time of onset of sensory block is defined as time interval between end of local anesthetics injection and complete loss of sensation to pin prick in all four nerve distribution areas, and the duration of sensory block is defined as the time interval between onset of sensory block and reappearance of pinprick sensation in all four nerve distribution areas.
Time of onset of motor block | Intraoperatively
  Time of onset of motor block is defined as the time interval between the completion of local anesthetics injection and the inability of patient to move the elbow, wrist and fingers of the operating limb.
Degree of pain | 24 hours postoperatively
  Degree of pain will be recorded using numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). It will be assessed every 2 hours for 6 hours then every 4 hours for 24 hours postoperatively.
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated) will be recorded.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as local anesthetics systemic toxicity, PONV, hypotension, pneumothorax, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author